CLINICAL TRIAL: NCT04318353
Title: The Effect of Early Enteral Feeding on Neonatal Outcome After Gastrointestinal Tract Surgery
Brief Title: The Effect of Early Enteral Feeding on Neonates After GIT Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sandy Nashat Rezk Abaskharon, Principal investigator, Assiut University
Other Study IDs: EEF neonates after GIT surgery
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Post-Gastrointestinal Tract Surgery Malnutrition
Keywords: neonatal feeding; gastrointestinal tract surgery
MeSH Terms: interventions — Postoperative Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- early enteral feeding: start enteral feeding within 2 days postoperative
  Interventions: Other: early enteral feeding within 2 days postoperative
- control: start enteral feeding after 2 days postoperative according to clinician discretion based on clinical progress(ranging from 1-5 days after passage of flatus or stool.

INTERVENTIONS:
Other: early enteral feeding within 2 days postoperative — Enteral feeding within 2 days postoperative
  Groups: early enteral feeding

SUMMARY:
This study aims to evaluate the effect of early vs late enteral feeding after abdominal surgery on neonatal outcome after surgery, weight gain, length of hospital stay, time to reach full enteral feeding, time to pass first stool, surgical site infections, sepsis and electrolyte disturbances.

DETAILED DESCRIPTION:
There are a many reasons for gastrointestinal (GI) tract surgery and following surgery the aim is to efficiently establish infants on enteral feeds and wean them off of parenteral nutrition. Neonates may lose their body resources after surgery due to inadequate nutrient intake and undergoing long periods of fasting after surgery. Nil peroral (NPO)/nil by mouth has been the most commonly practiced convention in post-operative period. Misplaced fear of aspiration, prevent nausea, vomiting and anastomotic complications led to routine prescription of "NPO." The duration of postoperative fasting is variable but can range from 0 to 5 days depending on the operation. The ramiﬁcations of this period of fasting are not insigniﬁcant and may include prolonged length of stay, increased use of parenteral nutrition (PN), social effects and signiﬁcant costs to the health system.

Starvation leads to disuse atrophy of villi, decrease disaccharide activity, decreased intestinal mucosa mass, and loss of DNA of enterocyte. This malfunctioning enterocyte leads to increase the permeability of intestinal mucosa to antigen and macromolecules. This starvation-induced gut mucosal injury leads to decrease the production of Vitamin K due to the absence of normal colonic flora. This also leads to decreased growth factors and bile acid metabolism. This compounded effect of starved gut and abnormal colonic bacterial environment leads to colonization of pathological bacteria and might lead to sepsis and sequelae. In addition, starvation leads to decreased immune cells of intestine gut-associated lymphoid tissue. This decreased gut immunity leads to increased uptake of toxins and decreased immune response to foreign antigen. This leads to bacterial translocation Traditionally after abdominal surgery, presence of bowel sounds or passage of flatus or stools has been the clinical evidence of restoration of bowel activity and indicators for starting oral diet. Bowel sounds are poor markers of bowel function as uncoordinated and antegrade peristalsis can be heard as bowel sounds. Currently, there is no good marker for return of bowel sounds, and even in the presence of prolonged ileus, the bowel moves .

Cochrane reviews have shown no advantage in keeping patients "nil by mouth" following gastrointestinal surgery and support early commencement of enteral feeding .

In neonates and infants there are additional issues with delayed feeding including cholestatic jaundice, sepsis, delayed gut development, and metabolic disease. Early trophic feeds may improve recovery time by increasing gut blood flow, improving motility and limiting the impact of starvation on the structure of the gut and its ability to absorb nutrients. Early introduction of enteral nutrition improves intestinal adaptation, reducing the risk of intestinal failure-associated liver disease (IFALD).

ESPEN guidelines recommend early initiation of enteral feeding within 24 h after gastrointestinal surgery, but also state that it needs to be adapted according to the individual tolerance and type of surgery .

So this study aims to evaluate the effect of early vs late enteral feeding after abdominal surgery on neonatal outcome after surgery, weight gain, length of hospital stay, time to reach full enteral feeding, time to pass first stool, surgical site infections, sepsis and electrolyte disturbances and will include all neonates who undergoing abdominal surgery and admitted in neonatal intensive care unit in Assiut University Children Hospital for one year.

The study will include 2 groups group A :start enteral feeding within 2 days postoperative and group B :start enteral feeding after 2 days postoperative according to clinician discretion based on clinical progress(ranging from 1-5 days after passage of flatus or stool.

ELIGIBILITY:
Inclusion Criteria:

* All admitted neonates who undergo abdominal surgery

Exclusion Criteria:

* Neonates with no-abdominal surgery.
* Neonates on mechanical ventilation
* Neonates with other co-morbidities like sepsis, severe respiratory distress, intracranial hemorrhage, birth asphyxia, congenital heart diseases and multiple congenital anomalies

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all neonates who undergoing abdominal surgery and admitted in neonatal intensive care unit in Assiut University Children Hospital for one year
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
weight gain | One year
  Follow up and record of weight after surgery every 24 hours and compaire the results between the two groups

SECONDARY OUTCOMES:
Length of hospital stay | One year
  Record the length of hospital stay for each patient
Time to reach full enteral feeding | One year
  Record the time to reach full enteral feeding for each patient and compaire the average time between the 2 groups
Time to pass first stool | One year
  Record the time to pass first stool and compair the average time between the 2 groups
surgical site infections | One year
  Observe the patients for signs of surgical site infection and record the number of patients who has surgical site infection in the groups
sepsis | One year
  Observe the patients for signs of sepsis and record the number of patients who has sepsis in the groups
electrolyte disturbances | One year
  Electrolytes measurment is routinely done for each surgical patient we will record the result in our study and take the average for each group for comparison

CONTACTS AND LOCATIONS:
Overall Officials: Azza A El Tayeb, MD, Study Director — Assiut University

REFERENCES:
- [Result] Andersen HK, Lewis SJ, Thomas S. Early enteral nutrition within 24h of colorectal surgery versus later commencement of feeding for postoperative complications. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD004080. doi: 10.1002/14651858.CD004080.pub2. PMID 17054196
- [Result] Weimann A, Braga M, Harsanyi L, Laviano A, Ljungqvist O, Soeters P; DGEM (German Society for Nutritional Medicine); Jauch KW, Kemen M, Hiesmayr JM, Horbach T, Kuse ER, Vestweber KH; ESPEN (European Society for Parenteral and Enteral Nutrition). ESPEN Guidelines on Enteral Nutrition: Surgery including organ transplantation. Clin Nutr. 2006 Apr;25(2):224-44. doi: 10.1016/j.clnu.2006.01.015. Epub 2006 May 15. PMID 16698152
- See also: Neonatal feeding: care and outcomes following gastrointestinal surgery. — http://www.infantjournal.co.uk/journal_article.html?RecordNumber=6936
- See also: Effects of Early Feeding Support on the Postoperative Weight Gain Status of Infants with Esophageal Atresia — http://ebcj.mums.ac.ir/article_7327.html
- See also: Have you passed gas yet? Time for a new approach to feeding patients post operatively. — https://www.google.com/url?sa=t&source=web&rct=j&url=https://med.virginia.edu/ginutrition/wp-content/uploads/sites/199/2015/11/SchulmanArticleOct-05.pdf&ved=2ahUKEwj5y9C2wqToAhXOVhUIHb0tDF4QFjAAegQIARAB&usg=AOvVaw0X3Fc2mO3vqzC8JaVFIQDo
- See also: Early feeding in tracheo esophageal fistula repair: Newer trends in post-operative care — http://www.medicinesjournal.com/archives/2016/vol1/issue2/1-2-31
- See also: Early enteral feeding following repair of gastroschisis is associated with shorter length of admission and better nutritional outcomes — http://www.jcnonweb.com/article.asp?issn=2249-4847;year=2017;volume=6;issue=4;spage=231;epage=235;aulast=Thompson